CLINICAL TRIAL: NCT02095366
Title: Intra Nasal Sufentanil Versus Intravenous Morphine for Acute Severe Traumatic Pain Analgesia in Emergency Setting. A Multicenter,Randomized,Controled, Comparative, Double Blinded Study
Brief Title: Intra Nasal Sufentanil Versus Intravenous Morphine for Acute Severe Traumatic Pain Analgesia in Emergency Setting
Acronym: ALGOFINE-2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Fondation Apicil (Other); SFMU (Unknown)
Responsible Party: Principal Investigator, AdministrateurDRC, Delegation de la recherche clinique et de l'innovation, University Hospital, Grenoble
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ALGOFINE-2
Record Dates: First submitted 2014-02-11; First posted 2014-03-24 (Estimated); Last update posted 2025-08-13 (Actual); Status verified 2017-12

CONDITIONS: Severe Traumatic Pain; Numeric Pain Rating Scale > 5 / 10
Keywords: Acute Pain; Traumatic Pain; Emergency setting; Prehospital setting; Analgesia; Intranasal device; Intra veinous injection; Sufentanil citrate; Morphine Sulfate
MeSH Terms: conditions — Acute Pain; Agnosia | interventions — Morphine; Sufentanil; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IN Sufentanil AND IV Placebo (Experimental): Patient receives silmutaneously intranasal sufentanil spray AND intraveinous placebo administration
  Interventions: Drug: Sufentanil; Drug: Placebo
- IV Morphine AND IN Placebo (Active Comparator): Patient receives silmutaneously intraveinous morphine administration AND intranasal placebo spray
  Interventions: Drug: Morphine; Drug: Placebo

INTERVENTIONS:
Drug: Morphine — Intravenous administration Patient receives simultaneously IV morphine administration and IN placebo spray.
  Pain is controlled by:
  * at 0 minute : Placebo IN (2 sprays, one spray in each nostril) + morphine IV 0,1mg/kg
  * at 10 minutes and if NPRS>3 : Placebo IN (1 spray) + morphine IV 0,05mg/kg
  * at 20 minutes and if NPRS>3: Pacebo (1 spray) + morphine IV 0,05mg/kg
  Arms: IV Morphine AND IN Placebo
Drug: Sufentanil — Intranasal spray with one spray, equivalent to an half-dose. Patient receives simultaneously IV placebo administration and IN sufentanil spray.
  Pain is controlled by:
  * at 0 minute : Sufentanil IN 0,3µg/kg (2 sprays, one spray in each nostril) + NaCl 0,9% IV
  * at 10 minutes and if NPRS>3 : Sufentanil IN 0,15µg/kg (1 spray) + NaCl 0,9% IV
  * at 20 minutes and if NPRS>3: Sufentanil IN 0,15µg/kg (1 spray) + NaCl 0,9% IV
  Arms: IN Sufentanil AND IV Placebo
Drug: Placebo — Intravenous administration Patient receives simultaneously IV placebo administration and IN sufentanil spray.
  Pain is controlled by:
  * at 0 minute : Sufentanil IN 0,3µg/kg (2 sprays, one spray in each nostril) + NaCl 0,9% IV
  * at 10 minutes and if NPRS>3 : Sufentanil IN 0,15µg/kg (1 spray) + NaCl 0,9% IV
  * at 20 minutes and if NPRS>3: Sufentanil IN 0,15µg/kg (1 spray) + NaCl 0,9% IV
  Other Names: saline solution; NaCl 0.9%
  Arms: IN Sufentanil AND IV Placebo
Drug: Placebo — Intranasal spray with one spray, equivalent to an half-dose. Patient receives simultaneously IV morphine administration and IN placebo spray.
  Pain is controlled by:
  * at 0 minute : Placebo IN (2 sprays, one spray in each nostril) + morphine IV 0,1mg/kg
  * at 10 minutes and if NPRS>3 : Placebo IN (1 spray) + morphine IV 0,05mg/kg
  * at 20 minutes and if NPRS>3: Pacebo (1 spray) + morphine IV 0,05mg/kg
  Other Names: saline solution; NaCl 0.9%
  Arms: IV Morphine AND IN Placebo

SUMMARY:
Intranasal (IN) administration of opiates is an appealing non-invasive way of treating acute traumatic pain in prehospital and Emergency departments (ED).

The investigators hypothesize that IN administration of Sufentanil is equal as compared with Intra veinous (IV) administration of Morphine wich is widely recommended in ED.

The investigators study is a multicentric, comparative, randomized, double-blind, double-placebo study, comparing quality of analgesia in both groups 30 minutes after first administration of opiates.

The investigators also asses side effects and patient satisfaction in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic pain
* Numeric Pain Rating Scale (NPRS) >5 /10
* Age between 18 and 75 years old

Exclusion Criteria:

* Medical pain (headache, chest pain,...)
* Respiratory, renal or hepatic insufficiency
* Drug addiction
* Medical or Chirurgical sinus history
* Oxygene saturation < 90%
* Systolic blood pressure < 90mmHg
* Head injury with a neurological Glasgow Coma Scale (GCS) < 14
* Opioid allergy
* Facial traumatism
* Patient unable do understand or assessing NPRS
* Opiates administration within 6 hours before admission

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2013-08-02 (Actual); Primary Completion 2016-04-10 (Actual); Study Completion 2016-06-30 (Actual)

PRIMARY OUTCOMES:
Efficiency of Analgesia | 30 minutes
  Patient self-assessed pain intensity using Numeric Pain Rating Scale (0 to 10). 30 minutes after the first opiate administration.

SECONDARY OUTCOMES:
Opioid-related side effects | 10 minutes
  Sedation Score, Breathing Rate, Oxygen Saturation, Arterial Blood Pressure, Heart rate, Nasal Ulceration.
  Proportion of patients having opioid-related side effects.
Efficiency of Analgesia | Every 10 minutes
  Patient self-assessed pain intensity using Numeric Pain Rating Scale (0 to 10). 10 minutes and 20 minutes after the first opiate administration.
Patient Satisfaction | 40 min
Specific Analysis for the pre hospital setting group: Efficiency of Analgesia | Every 10 minutes
  Patient self-assessed pain intensity, using Numeric Pain Rating Scale (0 to 10) at 10, 20 and 30 min after the first opiate administration

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - Emergency Department - Hospital Albertville, Albertville
  - Emergency Department - Hospital Annecy, Annecy
  - Emergency Department - Hospital Chambéry, Chambéry
  - Emergency Department - University Hospital of Grenoble, Grenoble
  - Emergency Department - Hospital Saint Jean de Maurienne, Saint-Jean-de-Maurienne
  - Emergency Department - Hospital Voiron, Voiron

REFERENCES:
- [Result] Blancher M, Maignan M, Clape C, Quesada JL, Collomb-Muret R, Albasini F, Ageron FX, Fey S, Wuyts A, Banihachemi JJ, Bertrand B, Lehmann A, Bollart C, Debaty G, Briot R, Viglino D. Intranasal sufentanil versus intravenous morphine for acute severe trauma pain: A double-blind randomized non-inferiority study. PLoS Med. 2019 Jul 16;16(7):e1002849. doi: 10.1371/journal.pmed.1002849. eCollection 2019 Jul. PMID 31310600